CLINICAL TRIAL: NCT02112097
Title: ASIS for Enbrel in Plaque Psoriasis
Acronym: ASISinPP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ASIS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCTAR066986; R44AR066986 (Other Grant/Funding Number: NATIONAL INSTITUTE OF ARTHRITIS AND MUSCULOSKELETAL AND SKIN DISEASES)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Plaque Psoriasis.
Keywords: Plaque Psoriasis.; Subdermal bloodless space; Subdermal injection; Subcutaneous injection; Injectable electromyography needle; Electrical stimulation; MRI with Gadolinium
MeSH Terms: interventions — Gadolinium; Gadolinium DTPA; Etanercept

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- For Left Upper Arm (Experimental): For Left Upper Arm Total Persistent % subdermally, For Left Upper Arm Total Persistent % subcutaneously, and For Left Upper Arm Relative Prolongation Ability Score.
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- For Right Upper Arm (Experimental): For Right Upper Arm Total Persistent % subdermally, For Left Upper Arm Total Persistent % subcutaneously, and For Left Upper Arm Relative Prolongation Ability Score.
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Interventions: Drug: Gadolinium
- sPGA 50 n(%) (Experimental): sPGA 50 n(%) as Efficacy of Enbrel subcutaneously at Week 12, Efficacy of Enbrel subcutaneously at Week 24, and Efficacy of Enbrel subcutaneously at Week 36 vs. Efficacy of Enbrel subdermally at Week 12, Efficacy of Enbrel subdermally at Week 24, and Efficacy of Enbrel subdermally at Week 36. sPGA 50 n(%) "clear" or "minimal" is the % of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and % of patients with a reduction of PASI of at least 50% from baseline.
  Interventions: Drug: Efficacy of Enbrel subcutaneously at Week 12; Drug: Efficacy of Enbrel subcutaneously at Week 24; Drug: Efficacy of Enbrel subcutaneously at Week 36; Drug: Efficacy of Enbrel subdermally at Week 12; Drug: Efficacy of Enbrel subdermally at Week 24; Drug: Efficacy of Enbrel subdermally at Week 36
- PASI 75 n(%) (Experimental): PASI 75 n(%)
  Response to treatment defined as the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI, as PASI 75 n(%) subcutaneously at Week 12, PASI 75 n(%) subcutaneously at Week 24, and PASI 75 n(%) subcutaneously at Week 36 vs. PASI 75 n(%) subdermally at Week 12, PASI 75 n(%) subdermally at Week 24, and PASI 75 n(%) subdermally at Week 36.
  Interventions: Drug: PASI 75 n(%) subcutaneously at Week 12; Drug: PASI 75 n(%) subcutaneously at Week 24; Drug: PASI 75 n(%) subcutaneously at Week 36; Drug: PASI 75 n(%) subdermally at Week 12; Drug: PASI 75 n(%) subdermally at Week 24; Drug: PASI 75 n(%) subdermally at Week 36
- Adverse Injection site reactions (Experimental): Injection site reactions as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Heart failure (Experimental): Heart failure as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions Allergic Reactions (Experimental): Allergic Reactions as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions Blood/low blood counts (Experimental): Blood problems/low blood counts as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Nervous system (Experimental): Nervous system problems, such as multiple sclerosis, seizures, or inflammation of the nerves of the eyes, as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Infections (Experimental): Infections (upper respiratory infection, pyelonephritis, bronchitis, septic osteomyelitis, wound infection, pneumonia, foot abscess, leg ulcer), as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Malignancies (Experimental): Malignancies (lymphoma, basal & squamous skin cancer, non-cutaneous solid tumor, & Wegener's granulomatosis), as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Immunogenicity (Experimental): Immunogenicity as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36
- Adverse Reactions with Autoantibodies (Experimental): Autoantibodies, Lupus-like syndrome, autoimmune hepatitis, as Adverse Reactions of Enbrel subcutaneously vs. Adverse Reactions of Enbrel subdermally at Week 36.
  Interventions: Drug: Adverse Reactions of Enbrel subcutaneously; Drug: Adverse Reactions of Enbrel subdermally at Week 36

INTERVENTIONS:
Drug: Gadolinium — For Left Upper Arm Total Persistent % subdermally, on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm
Drug: Gadolinium — For Left Upper Arm Total Persistent % subcutaneously, on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Gadolinium Magnevist® (gadopentetate dimeglumine)
  .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm
Drug: Gadolinium — For Left Upper Arm Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium subcutaneously on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm
Drug: Efficacy of Enbrel subcutaneously at Week 12 — sPGA 50 n(%) as Efficacy of Enbrel subcutaneously at Week 12, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: Efficacy of Enbrel subcutaneously at Week 24 — sPGA 50 n(%) as Efficacy of Enbrel subcutaneously at Week 24, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: Efficacy of Enbrel subcutaneously at Week 36 — sPGA 50 n(%) as Efficacy of Enbrel subcutaneously at Week 36, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: Efficacy of Enbrel subdermally at Week 12 — sPGA 50 n(%) as Efficacy of Enbrel subdermally at Week 12, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: Efficacy of Enbrel subdermally at Week 24 — sPGA 50 n(%) as Efficacy of Enbrel subdermally at Week 24, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: Efficacy of Enbrel subdermally at Week 36 — sPGA 50 n(%) as Efficacy of Enbrel subdermally at Week 36, in terms of Proportion of patients who achieve a score of "clear" or "minimal" by the Static Physician Global Assessment (sPGA) and the proportion of patients with a reduction of PASI of at least 50% from baseline.
  The sPGA is a 6-category scale ranging from "5 = severe" to "0 = none" indicating the physician's overall assessment of the psoriasis severity focusing on indurations, erythema, and scaling. Treatment success of "clear" or "minimal" consists of none or minimal elevation in plaque, up to faint red coloration in erythema, and none or minimal fine scale over < 5% of the plaque.
  Other Names: Enbrel (etanercept)
  Arms: sPGA 50 n(%)
Drug: PASI 75 n(%) subcutaneously at Week 12 — PASI 75 n(%) as Efficacy of Enbrel subcutaneously at Week 12, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: PASI 75 n(%) subcutaneously at Week 24 — PASI 75 n(%) as Efficacy of Enbrel subcutaneously at Week 24, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: PASI 75 n(%) subcutaneously at Week 36 — PASI 75 n(%) as Efficacy of Enbrel subcutaneously at Week 36, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: PASI 75 n(%) subdermally at Week 12 — PASI 75 n(%) as Efficacy of Enbrel subdermally at Week 12, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: PASI 75 n(%) subdermally at Week 24 — PASI 75 n(%) as Efficacy of Enbrel subdermally at Week 24, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: PASI 75 n(%) subdermally at Week 36 — PASI 75 n(%) as Efficacy of Enbrel subdermally at Week 36, in terms of the proportion of patients who achieved a reduction in score of at least 75% from baseline by the PASI.
  Other Names: Enbrel (etanercept)
  Arms: PASI 75 n(%)
Drug: Adverse Reactions of Enbrel subcutaneously — Adverse Reactions of Enbrel subcutaneously at Week 36, in number of Injection site reactions, Heart failure, Allergic Reactions, Blood problems/low blood counts, Nervous system, Infections, Malignancies, Immunogenicity, and Autoantibodies.
  Other Names: Enbrel (etanercept)
  Arms: Adverse Injection site reactions; Adverse Reactions Allergic Reactions; Adverse Reactions Blood/low blood counts; Adverse Reactions with Autoantibodies; Adverse Reactions with Heart failure; Adverse Reactions with Immunogenicity; Adverse Reactions with Infections; Adverse Reactions with Malignancies; Adverse Reactions with Nervous system
Drug: Adverse Reactions of Enbrel subdermally at Week 36 — Adverse Reactions of Enbrel subdermally at Week 36, in number of Injection site reactions, Heart failure, Allergic Reactions, Blood problems/low blood counts, Nervous system, Infections, Malignancies, Immunogenicity, and Autoantibodies.
  Other Names: Enbrel (etanercept)
  Arms: Adverse Injection site reactions; Adverse Reactions Allergic Reactions; Adverse Reactions Blood/low blood counts; Adverse Reactions with Autoantibodies; Adverse Reactions with Heart failure; Adverse Reactions with Immunogenicity; Adverse Reactions with Infections; Adverse Reactions with Malignancies; Adverse Reactions with Nervous system
Drug: Gadolinium — For Right Upper Arm Total Persistent % subdermally, on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Gadolinium Magnevist® (gadopentetate dimeglumine) .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm
Drug: Gadolinium — For Right Upper Arm Total Persistent % subcutaneously, on MRI at 6 hrs, 12 hrs, and 24 hrs.
  Gadolinium Magnevist® (gadopentetate dimeglumine) .1cc/ diluted with .9cc normal saline subcutaneously for 30 patients, and subdermally with ASIS Device for 30 patients.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm
Drug: Gadolinium — For Right Upper Arm Relative Prolongation Ability Score or total Persistent % of Gadolinium subdermally over total Persistent % of Gadolinium subcutaneously on MRI.
  Other Names: Gadolinium Magnevist® (gadopentetate dimeglumine)
  Arms: For Left Upper Arm; For Right Upper Arm

SUMMARY:
AUTOMATIC SUBDERMAL INJECTOR SYSTEM (ASIS) Corporation has developed and patented the only automatic injection system for delivery of injectable products to the optimum spot, just outside of the fascia, which exists subdermally (between the skin and muscle) or interfascial (between the deeper muscles). ASIS device creates that bloodless space, enhancing Enbrel's efficacy and preventing unnecessary distant spread and adverse reactions. This space remains bloodless as long as the skin is lifted up or filled with an injectable product. Although ASIS device was initially designed to best administer BOTOX for such muscular conditions as Upper limb Spasticity, Cervical Dystonia, Chronic Migraine, Strabismus, Blepharospasm, and Primary Axillary Hyperhidrosis, the technology will also benefit other injectable products, including: GAMMAGARD for Primary Immunodeficiency (PI) and Insulin for Diabetics, etc.

DETAILED DESCRIPTION:
Over 6 months, Aim 1 will demonstrate that ASIS device consistently delivers an injectable product (e.g. Gadolinium) into that subdermal bloodless space. MRI is the most simple and logical imaging choice, preferred because with ultrasound, air is injected, which will dissipate too quickly out of bloodless space to allow measurements. Since there isn't a way to measure the level of Gadolinium within that subdermal bloodless space, at least the Prolongation of Gadolinium may be approximated by its greater or longer Persistent % on MRI. Also, since we can't assume that bloodless space for patients with a particular disease will behave the same way as normal patients or patients with different diseases, this approximation only works if the variables are minimized to the same particular skin affected by Plaque Psoriasis. Case in point, patients with Plaque Psoriasis tend to have thicker skin, so expectantly will have prolonged Gadolinium subcutaneously Persistent %, which may be very different from the other diseases and certainly from the skin of normal patients, while the Gadolinium subdermally Persistent % should remain the same. Therefore, the Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % subcutaneously, will be different and very specific for the particular skin affected by Plaque Psoriasis. However, they are valuable indicators that will help us modify the Enbrel dosage and duration to inject into that "unknown" subdermal space for Aim 2, from the "known" typical Enbrel dosage and duration for Plaque Psoriasis patients. For example, if Aim 1 found the Relative Prolongation Ability Score for the Plaque Psoriasis skin to be (2.00), then the typical subcutaneously Enbrel 50mg every 3 days, should be 25mg every 6 days subdermally.

Over 12 months, Aim 2 will again demonstrate the advantages of ASIS device injecting subdermally versus subcutaneously, but using Enbrel instead of Gadolinium on the particular skin affected by Plaque Psoriasis. Once we have shown ASIS device's consistent performance in Aim 1, then we may assume will deliver another product (Enbrel) into that bloodless space without the need to measure Enbrel's existent in that bloodless space. Using Enbrel instead of Gadolinium, we'll demonstrate the advantages of injecting subdermally over intramuscularly for the same affected skin sites in the same 60 adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria in general and for Gadolinium:
* Main Criteria for Inclusion: Eligible Ages: 12 Years to 65
* Genders Eligible for Study: Both
* Accepts Healthy Volunteers: Yes
* Must be outpatient, male or female, of any race, between 18 and 65 years of age.
* Must be able to understand the requirements of the study including maintaining a diary, and sign informed consent.
* Must be in good general health as determined by investigator.
* If female of childbearing potential, must have negative pregnancy test result at screening visit and practice reliable method of contraception
* Inclusion Criteria for Plaque Psoriasis in particular:
* Must have chronic moderate to severe plaque psoriasis and be candidates for systemic therapy or phototherapy.
* Must have psoriasis involving at least 10% of body surface and a minimum PASI score of 10.
* Patients are limited to low-moderate-strength topical corticosteroids in axillary, groin, and scalp regions.

Exclusion Criteria:

* Exclusion Criteria for Plaque Psoriasis in particular:
* Patients with guttate, erythrodermic, or pustular psoriasis and patients with severe infections within 4 weeks of screening are excluded from study.
* No concomitant major anti-psoriatic therapies are allowed during the study.
* Has chronic or recurrent infection, has been exposed to tuberculosis, has resided or traveled in areas of endemic tuberculosis or endemic mycoses, such as histoplasmosis, coccidioidomycosis, or blastomycosis; or has underlying conditions that may predispose them to infection such as advanced or poorly controlled diabetes

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Relative Prolongation Ability Score for Gadolinium subdermally injected. | 6 months
  Gadolinium will be injected with ASIS subdermally (30) or conventional subcutaneous (30) for 60 adult subjects with Plaque Psoriasis (involving at least 10% of body surface and a minimum Psoriasis Area & Severity Index (PASI) score of 10), just for the particular plaque skin area. The first MRI taken promptly after Gadolinium injection for each patient would be his or her reference of 100% Persistent, to which his or her subsequent MRI taken @ 6 hr, @ 12 hr, and @24hr later will be compared for Persistent %.This approximation can only work if the variables are minimized to the same population with Plaque Psoriasis, and the particular plaque skin area. The Relative Prolongation Ability Score or total Persistent % subdermally over total Persistent % subcutaneously, Plaque Psoriasis will be very valuable indicators for us to modify the Enbrel dosage and duration for testing with that "unknown" subdermal bloodless space in Aim 2.

SECONDARY OUTCOMES:
Efficacy of Enbrel subcutaneously vs. subdermally in Plaque Psoriasis. | 12 months
  Hypothetically, if that subdermal bloodless space in patients somehow failed to show prolongation of half-life for Gadolinium in Aim 1, we can still proceed with Aim 2, because Enbrel's Pharmacokinetics will be studied anyway, by following tumor necrosis factor, then comparing the Mean tumor necrosis factor receptor : Fc. However, the Pharmacokinetics of subdermally injected Enbrel will be just dependent on Enbrel's diffusion out of that subdermal bloodless space. Therefore, if Enbrel getting into the bloodstream becomes so severely inhibited, then we can just change the osmolality of Enbrel in the end. Response to treatment will be assessed after 3, 6 and 9 months of therapy, and defined as the patients who achieved a reduction in score of at least 75% from baseline by the PASI.8 Other therapeutic advantages of ASIS device subdermally over subcutaneously will also be studied by comparing the reduction of adverse reactions and injection site pain.

OTHER OUTCOMES:
Adverse Reactions of Enbrel subcutaneously vs. subdermally in Plaque Psoriasis | 12 months
  Adverse Reactions of Enbrel subcutaneously vs. subdermally:
  Heart failure, Allergic Reactions, Blood problems/low blood counts, Nervous system problems, such as multiple sclerosis, seizures, or inflammation of the nerves of the eyes, Infections (upper respiratory infection, pyelonephritis, bronchitis, septic osteomyelitis, wound infection, pneumonia, foot abscess, leg ulcer), Malignancies (lymphoma, basal & squamous skin cancer, non-cutaneous solid tumor, & Wegener's granulomatosis), Immunogenicity, Autoantibodies, Lupus-like syndrome, autoimmune hepatitis, and Injection site pain.

CONTACTS AND LOCATIONS:
Overall Officials: Li Nguyen, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM INC; Thanh Phung,, MD, Principal Investigator — AUTOMATIC SUBDERMAL INJECTOR SYSTEM, INC
Locations (1):
- Automatic Subdermal Injector System, Inc, Westminster, California, United States

REFERENCES:
- [Background] Fisher CJ Jr, Agosti JM, Opal SM, Lowry SF, Balk RA, Sadoff JC, Abraham E, Schein RM, Benjamin E. Treatment of septic shock with the tumor necrosis factor receptor:Fc fusion protein. The Soluble TNF Receptor Sepsis Study Group. N Engl J Med. 1996 Jun 27;334(26):1697-702. doi: 10.1056/NEJM199606273342603. PMID 8637514
- [Background] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107
- [Background] Bhutani T, Wong JW, Bebo BF, Armstrong AW. Access to health care in patients with psoriasis and psoriatic arthritis: data from National Psoriasis Foundation survey panels. JAMA Dermatol. 2013 Jun;149(6):717-21. doi: 10.1001/jamadermatol.2013.133. PMID 23783152
- [Background] Paonessa DF, Goldstein JC. Anatomy and physiology of head and neck infections (with emphasis on the fascia of the face and neck). Otolaryngol Clin North Am. 1976 Oct;9(3):561-80. No abstract available. PMID 980495
- [Background] Ramey DR, Fries JF, Singh G. The Health Assessment Questionnaire 1995 - Status and Review. In: Spilker B, ed. "Quality of Life and Pharmacoeconomics in Clinical Trials." 2nd ed. Philadelphia, PA. Lippincott-Raven 1996;227
- [Background] Enbrel (etanercept) Product Information http://pi.amgen.com/united_states/enbrel/derm/enbrel_pi
- [Background] GAMMAGARD LIQUID Comparison of Intravenous and Subcutaneous Administration in Primary Immunodeficiency Diseases (PID). http://www.clinicaltrials.gov/ct2/show/NCT00546871?term=Gammagard+subcutaneous&rank=5
- [Background] Magnevist (gadopentetate dimeglumine) Injection Product Information. http://bayerimaging.com/products/magnevist/safety-information_nsf.php
- See also: Click here for more information about this study ASIS for Enbrel in Plaque Psoriasis — http://www.asis-inc.com